CLINICAL TRIAL: NCT05563935
Title: A Study of Function-metabolism Coupling in Decision-making Confidence Neural Network of Obsessive-compulsive Disorder
Brief Title: Function-metabolism Coupling in Decision-making Confidence Neural Network of Obsessive-compulsive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2021-51
Record Dates: First submitted 2022-09-22; First posted 2022-10-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2021-09

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive-Compulsive Disorder; Case-control study; Repetitive transcranial magnetic stimulation; Decision-making confidence; Metabolism; Neural network; GABA
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OCD group (Active Comparator): OCD patients will receive rTMS treatment for 6 weeks.
  Interventions: Device: Repetitive transcranial magnetic stimulation
- HC group (No Intervention): Health control will not receive any treatment.

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation — The OCD group will receive rTMS treatment for 6 weeks. There are 5 rTMS treatments per week (Monday to Friday), and 30 rTMS treatments in total. Treatment is administered by Ma GPro X100 device (Maga Venture) with Cool-DB80 coil. Detailed parameters of rTMS: intensity of stimulus is 120% RMT; the frequency of trains is 1Hz and the number of pulses is 1; no intertrain intervals and the pulses number is 1000.
  Arms: OCD group

SUMMARY:
This study, a case-control study, aims to investigate the function-metabolism coupling in decision-making confidence neural network of obsessive-compulsive disorder.

DETAILED DESCRIPTION:
OCD shows various abnormalities in cognitive function. Decision-making confidence is a burgeoning research focus on cognitive abnormality of OCD. Gamma-aminobutyric acid (GABA) is a type of inhibitory amino acid. Some studies have indicated that GABA shows metabolic abnormality in OCD.

Repetitive transcranial magnetic stimulation (rTMS) is a safe and noninvasive treatment for OCD. This study intends to explore the differences of the function-metabolism coupling in decision-making confidence neural network between OCD and HC. And investigating the dynamic changes of the function-metabolism coupling after rTMS treatment (6 weeks) for OCD is another goal.

ELIGIBILITY:
Inclusion Criteria:

OCD group:

1. Age between 18 and 50 years.
2. Satisfied with the diagnostic criteria for OCD in DSM-V.
3. Taking medication or unmedication stably for 8 weeks or drug-naive.
4. YBOCS score ≥16.
5. Education level was limited to above middle school.
6. Has sufficient audiovisual skills to complete the necessary examinations for the study.
7. Right-handed (this criterion is for fMRI subjects only).
8. Subjects understood the study and signed informed consent.

HC group:

1. Match with the OCD group on age, gender, education years.
2. Unsatisfied with the diagnostic criteria for any mental disorder in DSM-V.
3. No history of taking psychotropic drugs.
4. No family genetic history of mental disorder.
5. Has sufficient audiovisual skills to complete the necessary examinations for the study.
6. Right-handed (this criterion is for fMRI subjects only).
7. Subjects understood the study and signed informed consent.

Exclusion Criteria:

OCD group:

1. Satisfied with the diagnostic criteria for a mental disorder in DSM-V other than OCD.
2. HAMD-17 score ≥ 17.
3. IQ < 70.
4. Obsessive-compulsive symptoms were too severe to participate in the experiment.
5. Hoarding symptom.
6. High risk of negative thought and suicide.
7. Severe central system or physical disease or drug abuse.
8. Pregnant women or women that getting ready for being pregnant and lactating.
9. With metal implants in the body, such as pacemakers, intracranial silver clips, metal dentures, arterial stents, arterial clips, joint metal fixation, or other metal implants, etc. (this criterion is for fMRI subjects only)

HC group:

1. High risk of negative thought and suicide.
2. HAMD-17 score ≥ 17.
3. IQ < 70.
4. Severe central system or physical disease or drug abuse.
5. Pregnant women or women that getting ready for being pregnant and lactating.
6. With metal implants in the body, such as pacemakers, intracranial silver clips, metal dentures, arterial stents, arterial clips, joint metal fixation, or other metal implants, etc. (this criterion is for fMRI subjects only)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Yale-Brown Obsessive-Compulsive Scale (YBOCS) | Change from Baseline at 6weeks
  YBOCS is compiled by Goodman in the United States and contains 10 items to assess the severity of obsessive thoughts and compulsive behavior. The scoring method adopts a five-point scale of 0-4 points, and the total score range is 0-40 points, which has good reliability and validity.

SECONDARY OUTCOMES:
Hamilton Depression Scale (HAMD-17) | Change from Baseline at 6weeks
  It is one of the most widely used examiner-rating depression scales, which contains 17 items. It is used to measure the severity of depression and its change in treatment. The total score range is 0-59, and a lower score means a better outcome.
Hamilton Anxiety Scale (HAMA-14) | Change from Baseline at 6weeks
  It is one of the most widely used examiner-rating anxiety scales, which contains 14 items. It is used to measure the severity of anxiety and its change in treatment. The scoring method adopts a five-point scale of 0-4 points. The total score range is 0-56 and a lower score means a better outcome.
Florida Obsessive Compulsive Inventory (FOCI) | Change from Baseline at 6weeks
  FOCI, a self-rating scale, is used to assess the severity of obsessive-compulsive symptoms within one month, which contains 20 items. The first 15 items are evaluated the symptoms by yes and no, and the last 5 items are evaluated the severity of symptoms on 0-4 five-point scale. The total score range is 0-20 and a lower score means a better outcome.
Obsessive Belief Questionnaire (OBQ-44) | Change from Baseline at 6weeks
  It is a self-rating scale to assess the severity of the obsessive belief, which contains 44 items. The scoring method adopts a seven-point scale of 1-7 points. The total score range is 44-308 and a lower score means a better outcome.
State-Trait Anxiety Inventory (STAI) | Change from Baseline at 6weeks
  It is one of the most widely used self-rating anxiety scales, which contains 40 items. The first 20 items are used to measure the state anxiety and the last 20 items are used to measure trait anxiety. The scoring method adopts a four-point scale of 1-4 points. Both the total score range of state anxiety and trait anxiety are 20-80 and a lower score means a better outcome.

OTHER OUTCOMES:
Decision-making confidence | Change from Baseline at 6weeks
  The decision-making confidence is measure by randomized dot motion (RDM) task with a self-reported confidence scale (1-4 points). And a lower score means a lower decision-making confidence.
The distribution and level of GABA in the brain | Change from Baseline at 6weeks
  Using the SPICE (an advanced MRI technology) to measure the distribution and level of gamma-aminobutyric acid (GABA) in the brain. The change of GABA metabolism will be observed during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Qing Fan, Doctor, Study Chair — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China